CLINICAL TRIAL: NCT02556385
Title: Effects of Repetitive Transcranial Magnetic Stimulation Based on Brain Activation During Language Performance in Stroke Patients With Non-fluent Aphasia: A Pilot Study
Brief Title: Effects of rTMS Based on Brain Activation During Language Performance in Stroke Patients With Non-fluent Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nam-Jong Paik, Professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-1507-308-006
Record Dates: First submitted 2015-09-13; First posted 2015-09-22 (Estimated); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Stroke; Aphasia
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- High frequency rTMS (Experimental): Most activated area from fNIRS with language task: Perileisional Broca's area
  Interventions: Device: High frequency rTMS
- Low Frequency rTMS (Active Comparator): Most activated area from fNIRS with language task: Contralesional homologs of Broca's area
  Interventions: Device: Low frequency rTMS

INTERVENTIONS:
Device: High frequency rTMS — Most activated area from fNIRS findings: Perileisional Broca's area, High frequency rTMS (10Hz), Number of total stimuli: 800, Location: perilesional Broca's area, Intensity: 100% of resting motor threshold, Coil orientation: tangential to scalp, in combination with speech therapy(35-40min) after each rTMS session, Daily 10 treatment session
  Arms: High frequency rTMS
Device: Low frequency rTMS — Most activated area from fNIRS findings: Contralesional homologs of Broca's area, Low frequency rTMS (1Hz), Number of total stimuli: 1200, Location: Contralesional homologs of Broca's area (Pars triangularis), Intensity: 90% of resting motor threshold, Coil orientation: tangential to scalp, in combination with speech therapy(35-40min) after each rTMS session, Daily 10 treatment session
  Arms: Low Frequency rTMS

SUMMARY:
The aim of this study is to assess the safety and clinical efficacy of high or low-frequency repetitive transcranial magnetic stimulation based on brain activation with functional near infrared spectroscopy in poststroke nonfluent aphasia patients.

DETAILED DESCRIPTION:
In poststsroke aphasia rehabilitation, repetitive transcranial stimulation (rTMS) studies aimed to reinforce the activity of the brain regions in the left hemisphere. This goal can be achieved by using an excitatory protocol to reactivate the perilesional area or inhibitory protocol to reduce activities in the contralesional area. However, most conventional rTMS studies employed an inhibitory low frequency protocol for the contralesional homologs of Broca's area.

In the present pilot study, investigators will perform functional near-infrared spectroscopy (fNIRS) prior to rTMS treatment for selection of the most appropriate application of stimulation. Stimulation site and protocol (high frequency or low frequency rTMS) will be determined by activation pattern from the fNIRS findings with language task in individual patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 yrs old
* Right-handed
* Radiologically confirmed left hemisphere stroke
* Fluent in Korean
* First ever stroke
* More than 1 year from stroke onset
* Non-fluent (motor-dominant) aphasia
* Written informed consent

Exclusion Criteria:

* Previous medical histories of stroke, cerebral vascular operation, seizure
* Patients with traumatic brain injury
* Unable to perform the language task
* Severe cognitive impairment (MMSE less than 16)
* Skin lesion in the stimulation site of scalp
* Metal implants in the body (cardiac pacemaker or aneurysm clip)
* Pregnancy, Breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
BNT (Boston naming test) | Before rTMS(baseline), after the completion of 10 session of treatment (rTMS+speech therapy), 2 weeks later after the completion of 10 session of treatment (rTMS+speech therapy)
  speech evaluation tool for measuring the confrontational word retrieval function

SECONDARY OUTCOMES:
WAB (Western aphasia battery) | Before rTMS(baseline), after the completion of 10 session of treatment (rTMS+speech therapy), 2 weeks later after the completion of 10 session of treatment (rTMS+speech therapy)
  speech evaluation tool for screening the presence, degree, and type of aphaisa
Laterality index (LI) | Before rTMS(baseline), after the completion of 10 session of treatment (rTMS+speech therapy), 2 weeks later after the completion of 10 session of treatment (rTMS+speech therapy)
  From fNIRS findings, LI=L-R/L+R (L and R represent maximum or mean left and Right hemisphereic Hbo values, respectively)

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Jong Paik, MD, PhD, Principal Investigator — Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seongnam, Korea
Locations (1):
- Department of Rehabilitation Medicine, Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seongnam-si, Korea, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided